CLINICAL TRIAL: NCT04003246
Title: Phase II Concurrent Durvalumab (MEDI4736) and Radiotherapy Followed by Consolidative Durvalumab (MEDI4736) for Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Concurrent Durvalumab and Radiotherapy for for Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Yuanyuan Zhang, MD, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1082
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer Stage III
Keywords: Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided

STUDY DESIGN:
Intervention Model Description: Patient registration Stage III non-small cell lung cancer Zubrod 0 or 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm: Therapeutic Intervention (Experimental): All subjects receive the same therapeutic intervention of 1500mg intravenous durvalumab once every 4 weeks while receiving a 60 Gy/30 Fraction course of thoracic radiotherapy. After radiotherapy is complete, subjects continue to receive 1500mg intravenous durvalumab once every 4 weeks for up to one year following the start of treatment.
  Interventions: Radiation: Thoracic RT and Durvalumab; Drug: Consolidative Durvalumab

INTERVENTIONS:
Radiation: Thoracic RT and Durvalumab — 1500mg every 4 weeks [Q4W] intravenous [IV], first dose within 3 days of RT initiation
  Other Names: 3D Conformal Radiation Therapy (3D-CRT); Intensity-Modulated Radiation Therapy (IMRT); Image-Guided Radiation Therapy (IGRT); Imfinzi
Drug: Consolidative Durvalumab — 1500mg every 4 weeks [Q4W] intravenous [IV] up to one year
  Other Names: Imfinzi

SUMMARY:
Single arm, Phase II trial of concurrent Durvalumab (MEDI 4736) and radiotherapy followed by consolidative Durvalumb (MEDI 4736) for Stage III Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
Immunotherapy has significantly improved the survival outcomes of patients with various cancer types including thoracic malignancies. In the PACIFIC study, patients with locally advanced NSCLC were randomized to the anti-PDL1 antibody durvalumab or placebo for up to 12 months after completion of concurrent chemoradiation. While NSCLC is typically considered relatively non-immunogenic, RT is thought to augment tumor immunogenicity(Iyengar & Gerber, 2013). The abscopal effect refers to the observation that the benefit seen in PACIFIC, along with the growing role of immunotherapy for the treatment advanced (stage IV) NSCLC, suggests that earlier exposure to durvalumab may improve outcomes and be well tolerated, thereby permitting de-escalation of therapy through removal of conventional chemotherapy from these regimens to a local area results in an antitumor effect distant to the radiation site.

Durvalumab (Imfimzi; MEDI4736; AstraZeneca) is a human monoclonal antibody of the immunoglobulin (Ig) G1 kappa subclass that inhibits binding of PD-L1 (B7-H1, CD274) to PD-1 (CD279) and CD80 (B7-1). MEDI4736 is composed of 2 identical heavy chains and 2 identical light chains, with an overall molecular weight of approximately 149 kDa. MEDI4736 contains a triple mutation in the constant domain of the Ig G1 heavy chain that reduces binding to complement protein C1q and the Fcγ receptors involved in triggering effector function. Durvlumab binds with high affinity and specificity to human PD-L1 and blocks its interaction with PD-1 and CD80

ELIGIBILITY:
Inclusion Criteria:

1.1 Pathologically (histologically or cytologically) proven diagnosis of NSCLC with, medically inoperable (or patients who refuse resection) stage IIIA or stage IIIB disease (AJCC 8th edition);

1.1.1 Inoperable Stage IIIA disease is defined by multiple and/or bulky N2 mediastinal lymph nodes on computed tomography (CT) scan such that, in the opinion of the treating investigator, the patient was not a candidate for surgical resection.

1.1.2 N2 disease must have been documented by biopsy, or at a minimum by fluorodeoxyglucose positron emission tomography (PET) or CT if nodes were more than 2 cm in short axis diameter.

1.1.3 T4 disease is often considered resectable at the discretion of a thoracic surgeon. Patients with T4N0 or T4N1 disease can be enrolled if their case is reviewed by a thoracic surgeon and felt to be unresectable or if they are either medically inoperable or refuse surgery.

1.1.4 Stage IIIB patients have N3 or T4N2 status. N3 status must have been documented by the presence of a contralateral (to the primary tumor) mediastinal lymph node or supraclavicular or scalene lymph node proven by biopsy, or at a minimum by fluorodeoxyglucose uptake on PET or more than 2 cm in short axis diameter on CT scan. Patients with disease extending into the cervical region (defined as disease extending above cricoid cartilage) are not eligible.

1.2 Appropriate stage for study entry based on the following diagnostic workup:

1.2.1 History/physical examination, including documentation of height, weight and vital signs, within 30 days prior to registration;

1.2.2 CT scan with IV contrast (CT scan without contrast acceptable if IV contrast is medically contraindicated) of the lung and upper abdomen through the adrenal glands within 60 days prior to registration (recommended within 30 days prior to registration);

1.2.3 MRI of the brain with contrast (or CT with contrast if MRI is medically contraindicated) within 60 days prior to registration; note: the use of intravenous contrast is required for the MRI or CT (unless medically contra-indicated).

1.2.4 Whole-body FDG-PET/CT within 60 days prior to registration;

1.3 Age ≥ 18 years;

1.4 Life expectancy ≥ 12 weeks

1.5 Zubrod Performance Status of 0-1 within 30 days prior to registration;

1.6 Adequate respiratory function within 180 days prior to registration defined as follows: FEV1 > 1.2 liters; DLCO ≥ 50% predicted;

1.7 Patients with post-obstructive pneumonia are eligible provided they no longer require intravenous antibiotics at registration;

1.8 Patients with a pleural effusion that is transudative, cytologically negative and non-bloody, are eligible if the radiation oncologist feels the tumor can be encompassed within a reasonable field of radiotherapy; if pleural fluid is too small a volume to effectively sample by thoracentesis and does not show increased metabolic activity on CT/PET imaging, the patient will be remain eligible.

1.9 Adequate organ and marrow function as defined below

1.9.1 Absolute neutrophil count >1.5 × 10^9/L

1.9.2 Platelet count >100 × 10^9/L

1.9.3 Baseline or post-transfusion Hemoglobin ≥9.0 g/dL

1.9.4 Serum bilirubin≤ 1.5x upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.

1.9.5 Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN.

1.9.6 Measured creatinine clearance (CL) >40 mL/min or calculated CL >40 mL/min as determined by Cockcroft-Gault (using actual body weight);

Males:

Creatinine CL = (Weight (kg) × (140 - Age)) / ((mL/min) 72 × serum creatinine (mg/dL))

Females:

Creatinine CL = (Weight (kg) × (140 - Age) × 0.85) / ((mL/min) 72 × serum creatinine (mg/dL))

1.10 Negative serum pregnancy test within three days prior to registration for women of childbearing potential.

1.11 Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

1.11.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

1.11.2 Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

1.12 Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

2.1 Definitive clinical or radiologic evidence of metastatic disease;

2.2 Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.

2.3 Current invasive malignancy (except non-melanomatous skin cancer, localized bladder and prostate cancer). Carcinoma in situ of the breast, oral cavity, or cervix are permissible regardless of timing;

2.4 Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields. For example, patients with prior breast radiotherapy treatments would likely be excluded;

2.5 Prior systemic treatment with chemotherapy, targeted therapy or an anti-PD-1, anti-PD-L1 including durvalumab, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways for locally advanced NSCLC. Prior chemotherapy and/or targeted therapy as adjuvant or neoadjuvant therapy for earlier-stage lung cancer is permitted as long as it was completed ≥6 months prior to enrollment. No prior anti-PD-1, anti-PD-L1 including durvalumab, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways is permitted.

2.6 A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease;

2.7 Severe, active co-morbidity defined as follows:

2.7.1 Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

2.7.2 Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone

2.7.3 Active infection including tuberculosis, hepatitis B, hepatitis C.

2.7.4 History of allogenic organ transplantation.

2.7.5 History of symptomatic or previously established interstitial lung disease;

2.7.6 History of severe hypersensitivity reaction to any monoclonal antibody or allergy to study drug components;

2.7.7 Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

2.8 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.

2.9 Pregnancy, nursing females, or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

2.10 Patients whose radiation treatment plans are likely to encompass a volume of whole lung receiving ≥ 35% of lung volume. V20s up to 37% will be permitted and viewed as a minor deviation, provided that the treating radiation oncologist believes this level of exposure is within patient tolerance.

2.11 Planned radiation cardiac dose V50 >25%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Zhang, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm: Therapeutic Intervention
Started | 10
Thoracic RT and Durvalumab | 10
Consolidative Durvalumab | 9
Completed | 1
Not Completed | 9
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 10
Age, Customized [Median (Full Range); unit: years]
  Median Age | 65.5 [56 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Black/African American | 1
  Non-Hispanic | 7
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 10
ECOG Performance Status [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out of work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  4: Completely disabled; cannot carry on any selfcare totally confined to bed or chair.
  5: Dead
  Participants
    0 | 2
    1 | 8
Smoking Status [Count of Participants; unit: Participants]
  Current | 2
  Former | 8

OUTCOME MEASURES:

1. Primary Outcome: 12-Month Progression-free Survival (PFS) Time
Description: To determine the 12-month progression-free survival (PFS) for Stage III non-small cell lung cancer patients treated with concurrent durvalumab and radiotherapy followed by consolidative durvalumab. PFS rate is based on an assessment by an investigator according to RECIST 1.1 criteria; PFS is defined as the time from the study enrollment to documented progressive disease or death due to any cause, whichever occurs first.
Time Frame: Twelve months from the study enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 10
days | 208 [0 to 365]

2. Secondary Outcome: Safety and Tolerability
Description: To assess the safety and tolerability of concurrent durvalumab and radiotherapy compared to historical data from patients treated with standard of care chemo-radiation using adverse event according to CTCAE V.5
Time Frame: 4 years from study enrollment
Measure: Number; unit: Grade 3 or higher adverse events
Units Other Than Participants: Grade 3 or higher adverse events
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 10
Number analyzed (Grade 3 or higher adverse events) | 22
Grade 3 or higher adverse events
  Treatment-related | 15
  Not treatment-related | 7

3. Secondary Outcome: Overall Survival
Description: To determine the overall survival (OS) defined as the time from study enrollment to death due to any cause
Time Frame: Up to 4 years (1461 days) from study enrollment
Population: Active, living participants and participants that have experienced death due to any cause.
Measure: Mean (Full Range); unit: days
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 10
days | 486 [0 to 1460]

4. Secondary Outcome: Distant Metastases Free Survival Time
Description: Time from study enrollment to any new distant lesion.
Time Frame: From date of study enrollment until the date of first documented new distant lesion or date of death from any cause, whichever came first, assessed to the end of the study (approximately 55 months).
Population: Active patients without demonstrated distant metastasis, patients with any distant metastatic new lesion, and deceased patients that were on the study.
Measure: Mean (Full Range); unit: days
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 10
days | 501 [0 to 1677]

5. Secondary Outcome: Local and Regional Control Time
Description: The time from the study enrollment to any local and regional lesion.
Time Frame: From date of study enrollment until the date of first documented local and regional lesion, assessed to the end of the study (approximately 55 months).
Population: Active participants and all previous patients with demonstrated new local and regional lesions.
Measure: Mean (Full Range); unit: days
Arm/Group | Single Arm: Therapeutic Intervention
Number analyzed (Participants) | 4
days | 457 [0 to 1677]

ADVERSE EVENTS:
Time Frame: Adverse have been collected from baseline until death of the patient or end of the study (approximately 4 years and 7 months). Adverse events were collected weekly during the concurrent phase (up to 6 weeks after enrollment), then monthly during the consolidative phase (up to 1 year after beginning the consolidative phase). Then, adverse events were collected every 3 months until 2 years post concurrent treatment. After year 3, adverse events were collected every 6 months until end of study.
Description: Adverse events are not divided into arms for concurrent vs consolidative durvalumab as all patients were prescribed the same treatment, and the aim of the study was not to separate the two factors.
Arm/Group | Single Arm: Therapeutic Intervention
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Therapeutic Intervention (N=10)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Therapeutic Intervention (N=10)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 4 (4)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Ear and labyrinth disorders - Other, ear discharge (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema Limbs (General disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (11)
Fever (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders - Other, dark stools, blood in stools (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, heat intolerance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, cold intolerance (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (5)
Investigations - Other, Iron decreased (Investigations) | 1 (1)
Investigations - Other, Neutrophil increased (Investigations) | 2 (2)
Investigations - Other, creatinine decreased (Investigations) | 4 (4)
Investigations - Other, T3 total decreased (Investigations) | 1 (2)
Investigations - Other, cortisol decreased (Investigations) | 1 (1)
Investigations - Other, ferritin increased (Investigations) | 1 (1)
Investigations - Other, free T4 increased (Investigations) | 1 (1)
Investigations - Other, TSH decreased (Investigations) | 1 (1)
Investigations - Other, phosphorus decreased (Investigations) | 1 (1)
Investigations - Other, ACTH decreased (Investigations) | 2 (2)
Investigations - Other, ALT decreased (Investigations) | 1 (1)
Investigations - Other, AST decreased (Investigations) | 1 (1)
Investigations - Other, BUN increased (Investigations) | 1 (1)
Investigations - Other, chloride decreased (Investigations) | 2 (4)
Investigations - Other, Eosinophils decreased (Investigations) | 1 (1)
Investigations - Other, free T3 decreased (Investigations) | 1 (2)
Investigations - Other, MCHC decreased (Investigations) | 1 (1)
Investigations - Other, Monocytes absolute increased (Investigations) | 1 (1)
Investigations - Other, MPV decreased (Investigations) | 1 (1)
Investigations - Other, platelet count increased (Investigations) | 2 (2)
Investigations - Other, RDW-CV increased (Investigations) | 1 (1)
Investigations - Other, Leukocyte count decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 3 (7)
Lung infection (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (17)
Metabolism and nutrition disorders - Other, polydipsia (Metabolism and nutrition disorders) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (6)
Non-cardiac chest pain (General disorders) | 5 (6)
Oral gingivitis (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, development of new lung nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, right upper lobe consolidation and traction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 3 (5)
Shingles (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, change in mole (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, oily and clammy skin (Skin and subcutaneous tissue disorders) | 1 (1)
Social circumstances - Other, food insecurity (Social circumstances) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Surgical and medical procedures - Other, chronic draining scrotal abscess (Surgical and medical procedures) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 8 (15)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5)
White blood cell decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04003246/Prot_SAP_000.pdf